CLINICAL TRIAL: NCT05049824
Title: Single Neodymium Magnet Anastomosis Procedure When Used to Create a Duodenal-Ileal Diversion for Subjects With Inadequate Weight Loss or Weight Regain Following Sleeve Gastrectomy
Brief Title: Procedure for Duodenal-Ileal Diversion for Patients With Weight Regain Following Sleeve Gastrectomy
Acronym: SNAP-PS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GI Windows, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIW 19-001
Record Dates: First submitted 2021-09-09; First posted 2021-09-20 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SFM Treatment Arm (Experimental): The subjects in this arm will receive the Self-Forming Magnet (SFM) System that will be used to create a duodenal-ileal diversion
  Interventions: Device: Self Forming Magnetic (SFM) Anastomosis System

INTERVENTIONS:
Device: Self Forming Magnetic (SFM) Anastomosis System — The SFM will be placed using an endoscope in the duodenum and laparoscopically into the ileum. A compression anastomosis will be created in each of the subjects and the diversion of enteral flow from the duodenum to ileum will create a metabolic effect that will induce weight loss and impact metabolic disease indicators

SUMMARY:
Study will monitor weight loss and metabolic indicators for subjects in single-center, single arm trial.

DETAILED DESCRIPTION:
Single-Center, Open-label Pilot Study to Evaluate the Safety and Effectiveness of the GI Windows Single Neodymium Magnet Anastomosis Procedure When Used to Create a Duodenal-Ileal Diversion for Subjects with Inadequate Weight Loss or Weight Regain Following Sleeve Gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age 22-65 years at screening
* Body mass index (BMI) ≥35 and ≤50
* Patient is ≥12 months but ≤ 60 months post sleeve gastrectomy who have inadequate weight loss or weight regain.
* Weight stable over 3-month period
* Negative H. pylori breath test
* Agrees to refrain from any type of additional bariatric or reconstructive surgery that would affect body weight for a duration of 2 years
* If female, subject must commit to not becoming pregnant for 24 months and agree to use contraception during this period
* Able to understand and sign informed consent documents.

Exclusion Criteria:

* Known or suspected allergy to nickel or titanium or nitinol
* Contraindication to general anesthesia
* Previous technical difficulty or failed endoscopy or contraindication to endoscopy of upper GI series
* Any previous major surgery on the stomach (excluding sleeve gastrectomy), duodenum, hepatobiliary tree (excluding gallbladder), pancreas, or right colon.
* Clinically significant findings during screening endoscopy at target region for compression anastomosis
* Uncontrolled hypertension
* Pre-existing severe comorbid cardio-respiratory disease
* History of type 1 diabetes or poorly controlled type 2 diabetes
* Abnormal liver biochemistry
* History of chronic gastrointestinal disease
* Specific genetic or hormonal cause of obesity
* Recent tobacco/nicotine product cessation (within 3 months prior)

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Weight Loss | 12 Months
  1. Weight loss measured as a percent of total body weight (TBW)

SECONDARY OUTCOMES:
Percent responders | 12 Months
  Percent of subjects losing at least 10% and 20% of baseline weight from baseline
Excess weight loss | 12 Months
  Mean change in Excess weight loss from baseline
Change in serum lipids | 12 Months
  Mean change in serum lipids from baseline
Change in blood pressure | 12 Months
  Mean change in blood pressure from baseline
Change in fasting glucose | 12 Months
  Mean change in fasting glucose in subjects with T2DM at baseline
Change in HbA1c | 12 Months
  Mean change in HbA1c in subjects with T2DM at baseline
Change in BMI | 12 Months
  Mean change in BMI from baseline
Change in Absolute Weight Loss | 12 Months
  Mean change in Absolute Weight Loss from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Roman Turro, MD, Principal Investigator — Gastroenterologist at Teknon Hospital
Locations (1):
- Centro Medico Teknon, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No